CLINICAL TRIAL: NCT06869798
Title: EFFECTIVENESS of ZINC AS an ADJUVANT to STANDARD THERAPY VERSUS STANDARD THERAPY ALONE in CHILDREN (5-10 YEARS) with MODERATE PERSISTENT ASTHMA
Brief Title: EFFECTIVENESS of ZINC AS an ADJUVANT to STANDARD THERAPY VERSUS STANDARD THERAPY ALONE in CHILDREN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Kaushal Shah, MD (Postgraduate Trainee), King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4141/REG/KEMU/22MD200024
Record Dates: First submitted 2022-06-22; First posted 2025-03-11 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Asthma in Children
Keywords: asthma in children; zinc; standard therapy; adjuvant
MeSH Terms: interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: Randamize clinical trial
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- n Group A will receive standard therapy along with oral zinc 20mg/day OD for 2 months (Experimental): n Group A will receive standard therapy along with oral zinc 20mg/day OD for 2 months., all the patients of both groups will be trained to maintain diary regarding questionnaire asked in asthma control test, followed up 4 weekly for 8 weeks
  Interventions: Drug: zinc sulphate
- n Group B will receive only Standard therapy. (Experimental): n Group B will receive only Standard therapy., all the patients of both groups will be trained to maintain diary regarding questionnaire asked in asthma control test, followed up 4 weekly for 8 weeks
  Interventions: Drug: zinc sulphate

INTERVENTIONS:
Drug: zinc sulphate — Group A (intervention) and Group B (non-intervention). The patients in Group A will receive standard therapy along with oral zinc 20mg/day OD for 2 months. While the patients in Group B will receive only Standard therapy.
  Then, all the patients of both groups will be trained to maintain diary regarding questionnaire asked in asthma control test, followed up 4 weekly for 8 weeks

SUMMARY:
The objective of this study is to compare the effectiveness of zinc as an adjuvant to standard therapy versus standard therapy alone in children with moderate persistent asthma, as assessed by the Asthma Control Test, in terms of:

1. Improvement in asthma control as measured by the Asthma Control Test (ACT) score.
2. Association of continuous variables (e.g., age and duration of illness) and categorical variables (e.g., sex) with asthma control.

HYPOTHESIS Zinc as an adjuvant to standard therapy is more effective than standard therapy alone in managing moderate persistent asthma in children.

DETAILED DESCRIPTION:
DESIGN OF STUDY This is a Randomized Controlled Trial. FOLLOW-UP PROTOCOL The patients will be evaluated at the beginning of the study and then followed up at four weeks and eight weeks after enrollment to assess the primary and secondary outcomes. PRIMARY OUTCOME To assess the improvement in asthma control based on the Asthma Control Test (ACT) score at 4 weeks and 8 weeks, respectively. SECONDARY OUTCOMES

To observe improvement in:

1. Asthma symptoms and medication use, as recorded in patient diaries.
2. Association of continuous variables (e.g., age, duration of illness) and categorical variables (e.g., sex) with asthma control. SAMPLE SIZE The Calculated sample size is 84 children (42 in each group: Intervention & Control arm). SAMPLING TECHNIQUE Simple random sampling using the lottery method. SAMPLE SELECTION INCLUSION CRITERIA

1. Children ( 5-10) years. 2. Either gender. 3.Patient diagnosed with asthma according to the operational definition 4.Child with acute exacerbation of asthma EXCLUSION CRITERIA

1. Children with diarrhea and malnutrition
2. Children with pulmonary disease(pneumonia, viral infection,cystic fibrosis)
3. Children with cardiovascular disease. . 4. Children already taking zinc supplementation. STUDY PROCEDURE After approval from the Institutional Review Board of King Edward Medical University, Mayo Hospital, Lahore, all children aged 5 to 10 years, of either gender, diagnosed with asthma as per the operational definition and fulfilling the inclusion criteria, presenting to the Department of Pediatric Medicine, Mayo Hospital, will be enrolled in this study. Verbal and informed written consent will be obtained from the parents/guardians of all participants. Data Collection & Randomization

1. Demographic data will be collected. 2. A detailed history regarding symptoms, onset, duration of illness, progression, medication, level of asthma control, and general physical and systemic examination will be conducted. 3. Patients with moderate persistent asthma will be identified. 4. Using simple random sampling (lottery method), patients will be assigned into two groups:

1. Group A (Intervention): Standard therapy + Oral Zinc 20mg/day OD for 2 months.
2. Group B (Control): Standard therapy only. Follow-Up & Assessment All patients will be trained to maintain a diary, documenting responses to the

   1. Asthma Control Test (ACT) and medication use.
   2. Patients will be followed up every 4 weeks for 8 weeks to evaluate asthma control and symptom improvement.

ELIGIBILITY:
Inclusion criteria

* Children ( 5-10) years.
* Either gender.
* Patient diagnosed with asthma according to the operational definition
* Child with acute exacerbation of asthma

Exclusion criteria

* Children with diarrhea and malnutrition
* Children with pulmonary disease(pneumonia, viral infection,cystic fibrosis)
* Children with cardiovascular disease. . • Children already taking zinc supplementation.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control Test (ACT) Scores From Baseline to 8 Weeks | Baseline, 4 weeks and 8 Weeks
  The effectiveness of zinc as an adjuvant to standard therapy in children with moderate persistent asthma will be assessed by changes in Asthma Control Test (ACT) scores.
  Scores will be categorized as:
  * Controlled- if ACT score ≥ 20
  * Partially Controlled- if ACT score is 16-19
  * Uncontrolled- if ACT score < 16
  The intervention will be considered effective if there is a statistically significant increase in ACT scores from baseline to 8 weeks.
Number of Emergency Visits Due to Asthma Exacerbation | Baseline, 4 weeks and 8 Weeks
  The total number of emergency visits due to asthma exacerbation will be recorded at each follow-up. A reduction in emergency visits will be considered indicative of effective treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Shabbir, MBBS,FCPS, Principal Investigator — Pediatrics Department King Edward Medical University Lahore
Locations (1):
- King Edward Medical University Lahore Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only the principal investigator, supervisor, and Institution Review Board will have access with patients data upon request

REFERENCES:
- [Background] King GG, James A, Harkness L, Wark PAB. Pathophysiology of severe asthma: We've only just started. Respirology. 2018 Mar;23(3):262-271. doi: 10.1111/resp.13251. Epub 2018 Jan 9. PMID 29316003
- [Background] Vijverberg SJH, Farzan N, Slob EMA, Neerincx AH, Maitland-van der Zee AH. Treatment response heterogeneity in asthma: the role of genetic variation. Expert Rev Respir Med. 2018 Jan;12(1):55-65. doi: 10.1080/17476348.2018.1403318. Epub 2017 Nov 21. PMID 29115880
- [Background] Siripornpanich S, Chongviriyaphan N, Manuyakorn W, Matangkasombut P. Zinc and vitamin C deficiencies associate with poor pulmonary function in children with persistent asthma. Asian Pac J Allergy Immunol. 2022 Jun;40(2):103-110. doi: 10.12932/AP-100620-0878. PMID 33274952
- [Background] Rerksuppaphol S, Rerksuppaphol L. Zinc Supplementation in Children with Asthma Exacerbation. Pediatr Rep. 2016 Dec 9;8(4):6685. doi: 10.4081/pr.2016.6685. eCollection 2016 Nov 17. PMID 28058103
- [Background] Khanbabaee G, Omidian A, Imanzadeh F, Adibeshgh F, Ashayeripanah M, Rezaei N. Serum level of zinc in asthmatic patients: a case-control study. Allergol Immunopathol (Madr). 2014 Jan-Feb;42(1):19-21. doi: 10.1016/j.aller.2012.07.008. Epub 2013 Jan 9. PMID 23312452
- [Background] Chen M, Sun Y, Wu Y. Lower circulating zinc and selenium levels are associated with an increased risk of asthma: evidence from a meta-analysis. Public Health Nutr. 2020 Jun;23(9):1555-1562. doi: 10.1017/S1368980019003021. Epub 2019 Nov 5. PMID 31685060